#### MEDICAL RECORD

INSTITUTE/CENTER: NCI

PRINCIPAL INVESTIGATOR: Azam Ghafoor, MD

STUDY NUMBER: 19C0127

**STUDY TITLE:** A Phase II Study of LMB-100 Followed by Pembrolizumab

in the Treatment of Adults with Mesothelin-Expressing Non- Squamous Non-Small Cell Lung Cancer

(NSCLC)

Cohort: Screening

Consent Version: 12/04/2019

## WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Azam Ghafoor, MD

Phone: 240-858-3289

Email: azam.ghafoor@nih.gov

## KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes the research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you to in making your decision about participating in this study. Additional information that may help you make a decision can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to join this study because you have a kind of lung cancer (NSCLC) that has not responded to prior standard therapies, such as chemotherapy and immunotherapy.

This consent form requests your permission for us to test if you are eligible for this study. Patients on the study will receive LMB-100 and pembrolizumab. LMB-100 is an investigational agent, meaning that it has not been approved by the US Food and Drug Administration to treat NSCLC. Pembrolizumab (Keytruda®), is approved in the USA and some other countries for many cancers including NSCLC. Pembrolizumab use in this study is investigational as it has not been approved in the combination with LMB-100. However, the FDA has given us permission to use pembrolizumab and LMB-100 in this study.

You may only participate in this study if your cancer is positive for mesothelin. With your consent, we will first obtain your tumor tissue to test for mesothelin. Mesothelin is a protein found on many different tumors, but in very few non-cancer cells. We are asking you to screen for this research study because you have NSCLC that might make mesothelin. If your cancer is positive for mesothelin, you will need to have tests and/or procedures to help your doctor verify

#### PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

File in Section 4: Protocol Consent (3)


whether you can participate. This is called screening. The exams, tests, and procedures you will have are part of the usual approach for your cancer. Most must be performed within 28 days before enrollment. These basic tests include blood tests, x-rays, and physical exams, etc. Other tests are described further on in this consent form. It is important that you read about them. These tests will not be performed if your tumor tissue tests negative for mesothelin.

You may not benefit from this screening evaluation.

You may choose not to be tested for eligibility or to have any other studies done.

You are free to stop participating in the trial at any time. If you decide to stop, the study doctor may ask you to agree to certain tests to make sure it is safe for you to stop.

The remaining document will now describe this research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

#### IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY IS THIS STUDY BEING DONE?

This is a research study. The purpose of this research study is to find out if pembrolizumab given after LMB-100 in patients whose NSCLC makes a protein called mesothelin. Mesothelin is found on many different tumors, but in very few non-cancer cells.

We are asking you to screen for this research study because you have NSCLC that might make mesothelin. You have either received or are unable to receive standard therapy. If you have received standard therapy, your disease has gotten worse after that treatment.

If your cancer cells do not make mesothelin, you will not be eligible for this study. Your blood, biopsy or other tissue may also be tested for other research purposes. However, this consent does not permit any additional studies that would test for genetics (i.e. tendency for diseases) that might be inherited from you by your children.

#### WHAT WILL HAPPEN DURING THE STUDY?

The following research tests will be performed to determine whether you are eligible for this trial:

Mesothelin testing: You must provide a sample tumor tissue for formal evaluation by the National Cancer Institute (NCI) Laboratory of Pathology. The tissue may be from a previous surgery or biopsy. If none is available, we will ask you to have a biopsy to provide a fresh sample. Your tumor tissue will be used to determine whether your tumor cells have

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (3)


mesothelin. If no tumor tissue is available for this evaluation and new biopsy is not possible then you will not be eligible for the trial. In addition, this sample of tumor tissue will be used for confirmation of diagnosis by the NCI Laboratory of Pathology.

If the Mesothelin testing research test shows that your tumor does not make mesothelin, then further screening tests will not be performed. Otherwise, screening will continue as described below with standard clinical tests that are normally used to assess your disease.

- ROS1 Immunohistochemistry: Your tumor sample will be tested to determine if ROS1 genetic mutations are present. If either of these mutations are present, your study doctor will discuss alternative therapies that you should try before participating in this study. If you have exhausted these treatment options already, you may be eligible to participate in this study.
- <u>LSI ALK</u> (anaplastic lymphoma kinase) Break Apart DNA FISH test: Your tumor sample will be tested to detect mutations in the ALK gene. If this mutation is present, your study doctor will discuss alternative therapies that you should try before participating in this study. If you have exhausted these treatment options already, you may be eligible to participate in this study.
- Oncomine: Your tumor sample will be tested to determine if EGFR, ALK or ROS1 genetic mutations are present. If any of these mutations are present, your study doctor will discuss alternative therapies that you should try before participating in this study. If you have exhausted these treatment options already, you may be eligible to participate in this study.
- <u>TruSight Oncology 500 Assay</u>: Your tumor sample will be tested to determine if EGFR, ALK or ROS1 genetic mutations are present. If any of these mutations are present, your study doctor will discuss alternative therapies that you should try before participating in this study. If you have exhausted these treatment options already, you may be eligible to participate in this study.

If any of the mutation research testing listed above shows that your tumor is positive for an EGFR, ALK or ROS1 mutation and your cancer is amenable to a target therapy that is more likely to cure your cancer than the treatment offered in this study, then further screening tests will not be performed. Otherwise, screening will continue as described below with standard clinical tests that are normally used to assess your disease.

You will need to supply a complete list of your current medications to the study doctor. This includes over-the-counter medications and herbal supplements. Some medications may interact adversely with the study drugs and it is important that your study doctor and prescribing physician be aware of any potential risks so that they can prescribe alternative medications as necessary. If you do not already do so, please carry a list of your medications at all times.


Laboratory results performed outside of the NIH may be accepted if they have been performed recently. Otherwise, you will need to come to NIH Clinical Center to have the following standard, clinical tests performed at the NIH to determine whether you are eligible for this trial, which include:

- Medical history and physical examination
- Routine blood and urine tests including pregnancy test in women who can have children. Pregnant women will not be allowed on study.
- CT scan and FDG PET/CT scan
- Electrocardiogram (ECG)
- Echocardiogram
- Blood for tumor markers (substances found in your blood that may be a sign of cancer)
- Test for tuberculosis infection

#### HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this screening and your cancer makes mesothelin, your involvement will last for as long as it takes us to know if you are eligible to participate on the treatment phase of the study. The length of time may range anywhere from 1-4 weeks. You may be required to come to NIH at least 1 time during screening. This visit may last anywhere from 1 to 3 days.

#### HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

As not all persons screened will be eligible for study therapy, up to 100 patients will be screened in this study in order to treat up to 23 subjects in the main study.

## WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

The following study procedures may have risks and cause discomfort while you participate on this study:

## **Blood Draws**

The risk for taking blood samples involves the withdrawal of between a few teaspoons and a halfcup of blood and the potential for bruising or infection that occurs with any blood draw.

Each time a blood sample is needed, a needle will be put into a vein in your arm (or into your central venous catheter, if you have one). You may feel pain when the needle goes through the skin. Other side effects associated with drawing your blood for blood tests may include infection, bruising, redness, discomfort or bleeding at the site of the needle stick, and possible lightheadedness and fainting.

# Echocardiogram:

An echocardiogram is used to evaluate the structure and function of your heart. It uses harmless sound waves which bounce off the heart structures as a series of echoes. The echoes are recorded on moving graph paper or a videotape. This test is unlikely to cause any discomfort.


#### TB Skin Test:

A TB or tuberculosis test determines if you have an infection called tuberculosis or if you have been exposed to the germ that causes tuberculosis. This test is done on the inside of your forearm. A small needle will be put just under your skin and a very small amount of fluid will be injected causing a little bump to rise.

# Electrocardiogram (ECG)

An electrocardiogram or ECG is a test that records the electrical activity of the heart. It is used to measure the rate and regularity of heartbeats as well as the size and position of the heart chambers, and the presence of any damage to the heart. For this test, you will be asked to lie down, and small patches that have an adhesive edge with a gel in the middle, called electrodes, will be placed on your arms, legs, and chest. The areas where the electrodes are placed will be cleaned and, if needed, some hair may be shaved or clipped to allow for better attachment of the electrodes. The adhesive from the patches may irritate your skin.

# **Tumor Biopsies and Effusions**

Tumor biopsies and tumor effusions: local anesthesia of the skin will be given prior to any tumor biopsy or effusion collection, in order to prevent painful sensations. However, you may still experience pain or discomfort at the biopsy site. Irritation, redness, swelling and/or bleeding may also occur. There is a risk of abnormal healing, fever, infection or of an allergic reaction to the anesthetic agent used to anesthetize the skin at the biopsy site. Once the sample has been obtained, a stitch may be used to close the wound and assist in healing. A separate consent will be provided to you if a new biopsy or effusion collection is needed.

## **Radiographic Tests**

MRI, CT, X-ray, Nuclear Medicine and PET scans are common standard imaging tests used in the diagnosis and monitoring of many diseases. Although these tests have been in use for many years, their potential long-term effects on the body are still being learned. The most common discomfort is the length of time a patient must lay still or flat while an X-ray or scan is being performed. Occasionally, a patient may become uncomfortable within the closed space of the scanners (claustrophobia), particularly during an MRI. If this occurs, cool air can be blown over you by a fan if desired or your doctor can order a medicine for you to help you relax during this scan. Keeping the room well lit can also reduce this claustrophobic feeling. If a contrast agent (the special dye) is given with the scan there is a small risk of having a reaction to the contrast. In the small group of patients who have a reaction, the most common symptoms are nausea, pain in the vein where the contrast was given, headache, a metallic or bitter taste in the mouth, and a warm or flushing feeling that lasts from 1-3 minutes. Rarely, these symptoms may require treatment. In very rare cases, people have had more severe allergic reactions that result in skin rashes, shortness of breath, wheezing, or lowering of the blood pressure. If you have had a reaction in the past, be sure to tell your doctor or nurse about it. The radiation dose you receive, if your scan includes the use of x-rays or radioactive chemicals, is within the safe limits defined by the NIH Radiation Safety Guidelines and is considered essential for your medical care. In some cases, you may require medicines to make you sleep so you can be still during the procedure. The risks from this sedation

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (3)


IRB NUMBER: 19C0127

IRB APPROVAL DATE: 01/28/2020

or anesthesia are dependent on the types of medication used. These risks will be fully explained to you prior to the procedure and a separate informed consent will be obtained for anesthesia.

An IV line may need to be inserted for administration of the contrast agent or anesthetic. This can cause pain at the site where the IV is placed and carries a small risk of bruising or infection.

#### **MRI Risks**

Magnetic resonance imaging (MRI) uses a strong magnetic field and radio waves to take pictures of the body. You may need to have an MRI completed if you are unable to have a CT scan for screening. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the MRI, you will lie on a table that can slide in and out of the cylinder. You will be in the scanner for about 45 minutes. You may be asked to lie still for up to 15 minutes at a time. While in the scanner you will hear loud knocking noises, and you will be fitted with earplugs or earmuffs to muffle the sound. You will be able to communicate with the MRI staff at all times during your scan, and you may ask to be moved out of the machine at any time. It is very important that you do not move your body inside the scanner.

People are at risk for injury from the MRI magnet if they have some kinds of metal in their body. It may be unsafe for you to have an MRI scan if you have pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metal prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, tattoos, an implanted delivery pump, or shrapnel fragments. Welders and metal workers may have small metal fragments in the eye. You will be screened for these conditions before having any MRI scan. If you have a question about metal in your body, you should inform the staff. You will be asked to complete an MRI screening form before each MRI scan you have.

In addition, all magnetic objects (like watches, coins, jewelry, and credit cards) must be removed before entering the MRI scan room.

People with fear of confined spaces may become anxious during an MRI. Those with back problems may have back pain or discomfort from lying in the scanner. The noise from the scanner is loud enough to damage hearing, especially in people who already have hearing loss. Everyone having a research MRI scan will be fitted with hearing protection. If the hearing protection comes loose during the scan, you should let us know right away.

There are no known long-term risks of MRI scans.

# Risks for gadolinium enhanced MRI scans:

#### **Procedure**

During part of the MRI you will receive gadolinium, a contrast agent, through an intravenous (iv) catheter. It will be done for both research and medical purposes.

#### **Risks**

The risks of an IV catheter include bleeding, infection, or inflammation of the skin and vein with pain and swelling.

Mild symptoms from gadolinium infusion occur in fewer than 1% of those who receive it and usually go away quickly. Mild symptoms may include coldness in the arm during the injection, a metallic taste, headache, and nausea. In an extremely small number, fewer than one in 300,000 people, more severe symptoms have been reported including shortness of breath, wheezing, hives, and lowering of blood pressure. You should not receive gadolinium if you previously had an allergic reaction to it. You will be asked about such allergic reactions before gadolinium is given.

People with kidney disease are at risk for a serious reaction to gadolinium contrast called "nephrogenic systemic fibrosis" which has resulted in a very small number of deaths. A blood test of your kidney function may be done within the month before an MRI scan with gadolinium contrast. You will not receive gadolinium for a research MRI scan if your kidney function is not normal or if you received gadolinium within the previous month.

Most of the gadolinium contrast leaves the body in the urine. However, the FDA recently issued a safety alert that indicates small amounts of gadolinium may remain in the body for months to years. The effects of the retained gadolinium are not clear. At this time, retained gadolinium has not been linked to health risks in people whose kidneys work well. The NIH IRB has approved the gadolinium schedule for this study.

Some types of gadolinium contrast drugs are less likely to remain than others. In this study, we will use the gadolinium contrast drugs that are less likely to remain.

Please tell your research team if you have had any MRI scans in the past 12 months. We will also give you additional information called a "Medication Guide." Upon request, we will give you individual information about retained gadolinium we see on your studies.

# What are the risks related to pregnancy?

If you are a woman who is breast feeding or pregnant, you may not take part in the screening if a biopsy sample is already available for mesothelin testing. If a sample is unavailable, a biopsy would need to be performed to obtain tumor tissue, however, the radiation and procedure risks associated with this may affect your baby or unborn child.

# What are the risks of radiation from being in the study?

This research study involves exposure to radiation from CT scans to help guide us during your tumor biopsy. Please note that this radiation exposure is not necessary for your medical care and is for research purposes only. The amount of radiation you will receive in this study for research is about 0.8 rem, which is within the NIH Radiation Safety Committee guidelines of 5 rem per year.

The average person in the United States receives a radiation exposure of 0.3 rem per year from natural sources, such as the sun, outer space, and the earth's air and soil. If you would like more information about radiation, please ask the investigator for a copy of the pamphlet, <u>An Introduction to Radiation for NIH Research Subjects.</u>

While there is no direct evidence that the amount of exposure received from participating in this study is harmful, there is indirect evidence it may not be completely safe. There may be a very slight increase in the risk of cancer.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (3)


Please tell your doctor if you have had any radiation exposure in the past year, either from other research studies or from medical tests or care at the NIH or other places/hospitals that use radiation. This way we can make sure that you will not receive too much radiation. Consider X-rays taken in radiology departments, cardiac catheterization, and fluoroscopy as well as nuclear medicine scans in which radioactive materials were injected into your body.

If you are pregnant or breast feeding, you will not be permitted to participate in this research study. It is best to avoid radiation exposure to unborn or nursing children since they are more sensitive to radiation than adults.

#### WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You may not benefit from being in this study.

However, if you are found to be eligible for the main study, your lesions could go away or get smaller if the main study treatment is effective. The treatment could also decrease some of your symptoms, including pain, that are caused by your tumor(s).

# Are there any potential benefits to others that might result from the study?

We do not know if you will receive personal medical benefit from allowing us to perform these screening tests. However, this testing may make you eligible for the main study.

If you become eligible for our treatment study and you choose to participate, you will be asked to review and sign an additional informed consent that discusses the main study details and risks of treatment.

#### WHAT OTHER OPTIONS ARE THERE FOR YOU?

You may choose not to be screened for eligibility or to have any other studies done.

#### **DISCUSSION OF FINDINGS**

#### New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### Return of research results

The results from the evaluations for this screening will be reported to you. You will be informed whether or not you are eligible for the main study at that time.

## EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your participation for the following reasons:

- if he/she believes that it is in your best interest
- if you are ineligible for the study
- if you become pregnant
- if new information shows that another treatment would be better for you
- if the study is stopped for any reason

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (3)


In any of the above situations, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the study, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to our collaborators or designated representatives.

# WILL YOUR SPECIMENS OR DATA BE SAVED FOR USE IN OTHER RESEARCH STUDIES?

As part of this screening, we are obtaining specimens and data from you. Tumor tissue taken from a prior biopsy will be used for mesothelin testing. If no tumor tissue is available, a new biopsy will be performed. We plan to use these data for studies going on right now, as well as studies in the future.

We may share your specimens and data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or industry sponsors of research. We may also put your research data in a large database for broad sharing with the research community. These databases are commonly called data repositories. These data repositories might or might not be located at the NIH. If your individual research data is placed in one of these repositories, it will not contain information that can easily identify you and only qualified researchers will be able to look at your data. These researchers must receive prior approval from individuals or committees that monitor the use of the research information.

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your specimens and data. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, if the specimens and data has been shared already with other researchers, it might not be possible to withdraw.

### Please place your initials in the blank next to Yes or No for each of the questions below:

| My specimen | ns and data may be stored and used for future research as described above. |
|---|---|
| Yes | No |
| Initials | Initials |
| <i>J</i> 1 | ns and data may be shared with other researchers and used by these researchers for ch as described above. |
| Yes | No |
| Initials | Initials |

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)
File in Section 4: Protocol Consent (3)


## How Long Will Your Data be Stored by the NIH?

If you are eligible for the study, your data will be stored at NIH indefinitely.

# Risks of Storage and Sharing of Specimens and Data

When we store your tissue specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity by removing information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your data.

# COMPENSATION, REIMBURSEMENT, AND PAYMENT

### Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this screening.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

The NCI generally does not cover expenses during screening. If you are scheduled for and begin treatment on the main study, the NCI will cover the cost for some of your expenses. Someone will work with you to provide more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

## **CONFLICT OF INTEREST (COI)**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

NIH-2977 (4-17)
File in Section 4: Protocol Consent (3)


#### CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING.

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- 1. The National Cancer Institute (NCI) and other government agencies, like the Food and Drug Administration (FDA) and the Office for Human Research Protections, which are involved in keeping research safe for people.
- 2. National Institutes of Health Intramural Institutional Review Board

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens and data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

# **Certificate of Confidentiality**

To help us protect your privacy, the NIH Intramural Program has received a Certificate of Confidentiality (Certificate). With this certificate, researchers may not release or use data or information about you except in certain circumstances.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) File in Section 4: Protocol Consent (3)


The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical records we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your medical record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

### POLICY REGARDING RESEARCH-RELATED INJURIES

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# PROBLEMS OR QUESTIONS

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Dr. Azam Ghafoor (azam.ghafoor@nih.gov or 240-858-3289). You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

#### CONSENT DOCUMENT

Please keep a copy of this document in case you want to read it again.

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (3)


MEDICAL RECORD

CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

| Signature of Research Participant | Print Name of Research Participant | Date |
|---|---|---|
| about this study and have been given the to make research decisions on behalf of the | LAR) for an Adult Unable to Consent: I have exportunity to discuss it and to ask questions. It the adult participant unable to consent and have to information in the above consent was described pate in the study. | am legally authorize<br>the authority to provid |
| Signature of LAR | Print Name of LAR | Date |
| | ant: I have read the explanation about this stud<br>questions. I give permission for my child to take | |
| Signature of Parent/Guardian | Print Name of Parent/Guardian | Date |
| Signature of Parent/Guardian (as application) | Print Name of Parent/Guardian | Date |
| <b>Assent:</b> (Use this section only when this requires a separate assent form for this | s process is approved by an IRB for older minor population.) | s. Do not use if an IR |
| I have had this study explained to me in it, and I have had the chance to ask ques | a a way that I understand, I have been given the stions. I agree to take part in this study. | opportunity to discus |
| Assent of Minor: (as applicable) | | |
| Signature of Minor | Print Name of Minor | Date |
| <b>G</b> | | |
| Investigator: | | |
| _ | Print Name of Investigator | Date |

# MEDICAL RECORD

CONSENT TO PARTICIPATE IN AN NIH CLINICAL RESEARCH STUDY

| by the IRB for use as the basis of translation. | | |
|---|---|---|
| Witness: | | |
| Signature of Witness* | Print Name of Witness | Date |
| *NIH ADMINISTRATIVE SECTION TO INTERPRETER: | BE COMPLETED REGARDING T | HE USE OF AN |
| An interpreter, or other individual, who speather administration of informed consent and serve also serve as the witness. | | ~ ~ |
| An interpreter, or other individual, who speather administration of informed consent but did not providing interpretive support is: | | |

Witness to the oral short-form consent process only: This section is only required if you are doing the oral short-consent process with a non-English speaking subject and this English consent form has been approved

NIH-2977 (4-17) File in Section 4: Protocol Consent (3) 